CLINICAL TRIAL: NCT04523636
Title: Evaluation of Splinting in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: University of Maryland, Baltimore (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00075158
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injury Cervical; Splints
MeSH Terms: interventions — Splints

STUDY DESIGN:
Intervention Model Description: Each extremity was randomized to receive a custom or pre-fabricated resting hand splint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom Splint (Active Comparator): Custom Splint- Thermoplastic device fabricated by occupational therapist
  Interventions: Device: Splinting
- Prefabricated Splint (Active Comparator): Prefabricated Splint- Commercially available from Restorative Care of America, Inc (RCAI)
  Interventions: Device: Splinting

INTERVENTIONS:
Device: Splinting — Pre-fabricated or custom resting hand splints

SUMMARY:
This study compared pre-fabricated and custom resting hand splints among people who were in inpatient rehabilitation after a cervical spinal cord injury.

DETAILED DESCRIPTION:
This was randomized parallel group controlled clinical trial where arms, not patients were the unit of randomization. This trial was funded by the Craig H. Neilsen Allied Health Professional Development Award of the American Spinal Injury Association (ASIA). This research was conducted at a 32-bed spinal cord injury and multi-trauma rehabilitation unit in an urban center. Participants were recruited from an inpatient spinal cord injury rehabilitation unit. Eligible participants were 18 years or older and undergoing acute rehabilitation after a cervical spinal cord injury with hand function impairment, and the primary occupational therapist deemed splinting intervention was required. Each eligible extremity was randomized to receive a custom or pre-fabricated resting hand splint for night use.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury
* Inpatient Rehabilitation
* Limited hand function

Exclusion Criteria:

* Under 18
* Full hand function
* Orthopedic injury to hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in scores on The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP). | This assessment is completed within 5 days of initating the splinting intervention and within 3 days of discharge. Length of time between data collection was limited to 12 weeks.
  This test is a hand function assessment for spinal cord injury consisting of four domains- upper extremity strength, sensation, qualitative prehension, and quantitative prehension. Total scores for each upper extremity are calculated 0-116. Assessment of the Hand in Tetraplegia Using the Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP): Impairment versus Function.
  Kalsi-Ryan S, Curt A, Fehlings, MG and Verrier MC. Top Spinal Cord Inj Rehabil (2009); 14(4):34-46. - C

SECONDARY OUTCOMES:
Splint Perception Survey | This assessment was completed within 3 days of discharge and no more than 12 weeks after the intervention was initiated.
  This survey gathered participant perceptions via a 5 point Likert scale on the participant's perceptions of the splint's comfort and impact on function and hand position. Additionally, participants were asked to provide their perceptions on challenges to using the splint and advice to future therapists and patients considering splinting.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gorman, MD, Principal Investigator — University of Maryland, Baltimore; Paula Geigle, PhD, Principal Investigator — University of Maryland, Baltimore; Sara Frye, MS, Study Director — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of MD Rehabilitation & Orthopaedic Institute, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No